CLINICAL TRIAL: NCT01965444
Title: An Investigational, Non-significant Risk Study to Collect Data Needed to Analyze Readings Given by the SEM Scanner Point of Care 200 Series (SEM POC 200) and Its Ability to Detect Sub Epidermal Moisture.
Brief Title: A Test of the Investigational SEM Scanner
Status: Completed | Type: Observational
Sponsor: Bruin Biometrics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SEM200-001
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-10

CONDITIONS: Pressure Ulcers
Keywords: Sub-epidermal moisture; Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to establish required data for SEM Scanner analysis of the readings given by the SEM Scanner in the target patient population.. In order to better understand the data this non-invasive scanner provides a collection of data/readings is required to be collected in a certain population. This will help with clinical interpretation of the numbers and readings this device will provide.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are 18 years of age or older.
* Subject or health care proxy is willing and able to provide informed consent for enrollment.
* Subject is agreeable to having skin assessments, blanchability tests, and SEM Scanner readings performed daily at all anatomical sites for a duration of five (5) days, with photography as needed.
* Subject is admitted to an intensive Care Unit (ICU) and has an anticipated ICU course of 48 hours or greater.
* Subject is not Comfort Measures Only (CMO).
* Subject is anticipated to be bedridden for ore than 6 hours per day.
* All four (4) of the subject's anatomical sites in question (sternum, sacrum, left heel and right heel) are accessible for scanning (e.g., no cast or medical device present such that heels are not accessible).

Exclusion Criteria:

* Subject has broken skin or scar tissue at the sternum, sacrum, left heel or right heel.
* Subjects for whom the physical act of performing the inspections and measurements required in this study are contra-indicated, as determined by the principal investigator or attending physician.
* Subjects or legal representatives who are unable to understand the aims and objectives of the trial.
* Presence of any condition(s) which seriously compromise(s) the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
* Subject is pregnant.
* Subject is incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Units
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Descriptive statistic measurements | 5 day study period
  The endpoint for this study is the establishment of descriptive statistics around readings given by the SEM Scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Emhoff, MD, Principal Investigator — UMass Memorial Health
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States